CLINICAL TRIAL: NCT04168827
Title: Emotional and Social Impact on the Relatives of Hospitalized Children for Severe Trauma of 3 to 6 Months After the Intensive Care Unit Leaving
Brief Title: Emotional and Social Impact on the Relatives of Hospitalized Children for Severe Trauma
Acronym: RESPET
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190415; 2019-A01076-51 (Other: ID RCB number)
Record Dates: First submitted 2019-06-04; First posted 2019-11-19 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Severe Trauma
Keywords: Severe trauma; Post-traumatic stress; Anxiety; Depression; Intensive care
MeSH Terms: conditions — Wounds and Injuries; Anxiety Disorders; Depression | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Relatives of severe traumatized child: Relatives of a child who has been hospitalized in intensive care of Necker hospital following a severe trauma
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire completed by the parents of severe traumatized child, between 3 to 6 months after the leaving of the child out of intensive care unit

SUMMARY:
This research aims to study the occurrence of post-traumatic stress, anxiety or depression in the parents of a child who has been hospitalized in intensive care unit following a severe trauma.

DETAILED DESCRIPTION:
With nearly 25% of trauma deaths, trauma is one of the leading causes of death in the world for children aged 5 to 14 years. In children under 4, it is responsible for 6% of deaths.

Severe trauma is defined by an Abbreviated Injury Scale > 3 score in at least one anatomical region.

In case of multiple traumas, the Injury Severity Score is used to define severe polytrauma if it is > 15.

Cranial trauma is the most common lesion found in polytraumatized children and is present in 80% of cases.

Serious head trauma is defined as the existence of a cranial trauma in a patient whose Glasgow score is less than or equal to 8.

Severe trauma is a source of high mortality and severe disability in surviving children. Due to the context of sudden onset, a prolonged length of hospitalization in intensive care, as well as the occurrence of often severe sequelae, the severe trauma causes a real upheaval for the child's relatives.

In adults, the occurrence of post-traumatic stress, anxiety and depression is relatively well described in patients and relatives of patients who have been hospitalized in intensive care unit. However, there is currently no pediatric study focusing on this subject, apart from neonatology where the traumatological context remains exceptional.

This research aims to study the occurrence of post-traumatic stress, anxiety or depression in the parents of a child who has been hospitalized in intensive care unit following a severe trauma.

ELIGIBILITY:
Inclusion Criteria:

* Holder of the parental authority of a patient under 18 who has been hospitalized in the surgical intensive care unit of Necker University Hospital for severe trauma (Abbreviated Injury Scale greater than or equal to 3 in one of the anatomical regions) at the admission in the service and regardless of the ending of hospitalization.
* Holder of parental authority over 18 years.
* Holder of parental authority speaking French.

Exclusion Criteria:

* Holder of parental authority refusing to participate in the study, after submission of the information document.
* Holder of parental authority unable to answer the questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Holder of the parental authority of a patient under 18 who has been hospitalized in the surgical intensive care unit of Necker University Hospital for severe trauma (Abbreviated Injury Scale greater than or equal to 3 in one of the anatomical regions) at the admission in the service and regardless of the ending of hospitalization.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-12-09 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
Depression, post traumatic stress disorder, anxiety | 18 months
  Composite criterion considered positive if :
  The subject obtains a score greater than or equal to 13 in the Hospital Anxiety and Depression Scale questionnaire, thus defining a state of anxiety and depression. Hospital Anxiety and Depression Scale score range from 0 to 42 with higher scores indicating worse symptoms.
  and / or The subject obtains a score greater than or equal to 8 on one of the of the Hospital Anxiety and Depression Scale score. The Hospital Anxiety and Depression Scale score is separated in two section, one for Anxiety and one for depression. Each subscales range from 0 to 21 with higher scores indicating worse symptoms.
  and / or The subject obtains a score greater than or equal to 30 in the Impact of Event Scale Revised questionnaire defining high risk of presence of a post-traumatic stress disorder. The Impact of Event Scale Revised scores range from 0 to 88, with higher scores indicating worse symptoms.

SECONDARY OUTCOMES:
Socio-demographic analysis | 18 months
  A socio-demographic analysis of the population with data collected by a questionnaire focusing on :
  * Parent's age (in years)
  * The presence of a chronic disease (Yes/No)
  * The presence of psychiatric follow-up (Yes/No)
  * Taking antidepressant, neuroleptic or anxiolytic drugs (Yes/No)
  * Modification of marital status (Yes/No)
  * The presence of difficulties in the relationship with the spouse (Yes/No)
  * The evolution of professional status (No change / Loss of employment / Sickness leave / Decrease in professional activity)
  * The presence of financial difficulties (Yes/No)
Predictive factors for the occurrence of mental disorders | 18 months
  A search for predictive factors of the occurrence of a mental disorder will be conducted using the questionnaire and medical data from the child's file.
  Sub-group analyses will be carried out according to the results.
Feeling of hospitalization | 18 months
  The experience of relatives of hospitalization will be studied on the basis of the questionnaire focusing on :
  * Sufficient medical information by the team (Yes/No)
  * Suffering from the following situation:
    1. Visiting hours too restricted (Yes/No)
    2. Visits limited to parents (Yes/No)
    3. Insufficient availability of the medical team (Yes/No)
    4. Lack of availability of psychologists (Yes/No)
    5. Misunderstanding of the child's health problem (Yes/No)
  * Follow-up by a psychologist (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Meyer, Principal Investigator — Assistance Publique - Hôpitaux de Paris; Florian Prevost, Study Director — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No